CLINICAL TRIAL: NCT02030457
Title: A Randomized, Open-Label, 3-Period Crossover, Single-Dose Clinical Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Beclomethasone Dipropionate (160 and 320 mcg) Delivered Via Breath-Actuated Inhaler (BAI) and Metered-Dose Inhaler (MDI) in Healthy Adult Subjects
Brief Title: A Study to Investigate the Pharmacokinetics and Safety of Beclomethasone Dipropionate Administered by Breath-Actuated Inhaler and Metered-Dose Inhaler in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BDB-AS-101
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Treatment A: beclomethasone dipropionate BAI, 160 mcg - a single administration of 4 inhalations (40 mcg/inhalation)
  Interventions: Drug: Beclomethasone dipropionate BAI; Drug: Beclomethasone dipropionate MDI
- Treatment B (Experimental): Treatment B: beclomethasone dipropionate BAI, 320 mcg - a single administration of 4 inhalations (80 mcg/inhalation)
  Interventions: Drug: Beclomethasone dipropionate BAI; Drug: Beclomethasone dipropionate MDI
- Treatment C (Experimental): Treatment C: beclomethasone dipropionate MDI, 320 mcg - a single administration of 4 inhalations (80 mcg/inhalation)
  Interventions: Drug: Beclomethasone dipropionate BAI; Drug: Beclomethasone dipropionate MDI

INTERVENTIONS:
Drug: Beclomethasone dipropionate BAI — Breath Activated Inhaler (BAI)
Drug: Beclomethasone dipropionate MDI — Metered Dose Inhaler (MDI)

SUMMARY:
This study is designed to compare the systemic exposure of orally inhaled beclomethasone dipropionate inhalation aerosol delivered via BAI to that delivered via MDI.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a man or woman 18 through 45 years of age at the SV.
* The subject is assessed as being in good health based on a screening examination that includes medical history, physical examination (including a complete oropharyngeal examination), ECG assessment, and clinical laboratory results (ie, serum chemistry, hematology, and urinalysis).
* If female, subject is currently not pregnant, breast feeding, or attempting to become pregnant (for 30 days before the SV and throughout the duration of the study and for 30 days after subject's last visit), or is of non-childbearing potential, defined as any of the following:

  * pre-menarche
  * at least 1 year postmenopausal
  * surgically sterile (tubal ligation, bilateral oophorectomy, salpingectomy, or hysterectomy)
  * congenital sterility
  * diagnosed as infertile and not undergoing treatment to reverse infertility
  * or is of childbearing potential, has a negative serum pregnancy test, and is willing to commit to using a consistent and acceptable method of birth control as defined below for the duration of the study:
  * systemic contraception used for at least 1 month before the SV including birth control pills, transdermal patch (Ortho Evra®, Janssen Pharmaceuticals Inc., or equivalent), vaginal ring (NuvaRing®, Merck & Co., Inc., or equivalent), levonorgesterel implant (Norplant®, Population Council, or equivalent), or injectable progesterone (Depo-Provera®, Pfizer Inc., or equivalent)
  * double barrier methods (condoms, cervical cap, diaphragm, and vaginal contraceptive film with spermicide)
  * intrauterine device (IUD) with a low failure rate defined as less than 1% per year
  * monogamous with a vasectomized male partner or same-sex female partner
  * or is of childbearing potential and not sexually active, has a negative serum pregnancy test, and is willing to commit to using a consistent and acceptable method of birth control as defined above for the duration of the study, in the event the subject becomes sexually active.
  * If male, the subject is willing to commit to an acceptable method of birth control for the duration of the study, and for 3 months after dosing, or exclusively has same-sex partners.
* Subject is of normal body weight as evidenced by a BMI of at least 18 but no more than 30 kg/m2 (≥18 and ≤30 kg/m2), and has a body weight over 50 kg (>50 kg). The BMI is calculated as follows: weight (kg)/height2 (m).
* Subject does not have any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the subject at increased risk during the study.
* Other criteria may apply, please contact the investigator for more information.

Exclusion Criteria:

* Subject has clinically relevant abnormalities in clinical chemistry, hematology or any other laboratory variables.
* Subject has an irregular day/nighttime rhythm in daily living habits (eg, night work or repeated travels to places belonging to different time zones).
* Subject has been treated with any known cytochrome P450 3A4 (CYP3A4) inhibitor or inducers (eg, clarithromycin, ketoconazole, ritonavir, barbiturates, phenothiazines, cimetidine ) within 30 days before the Screening Visit (SV).
* Subject has been exposed to systemic corticosteroids (during the past 60 days) or intranasal/orally inhaled corticosteroids (during the past 30 days) for any indication, chronic or intermittent; or subject has an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
* Subject has used topical corticosteroids in concentrations in excess of 1% hydrocortisone or equivalent within 30 days before the SV; used a topical hydrocortisone or equivalent in any concentration covering greater than 20% of the body surface; or used any topical corticosteroids with an occlusive dressing; or has an underlying condition (as judged by the investigator) that can reasonably be expected to require treatment with such preparations during the course of the study.
* Subject has used any prohibited medication (see Section 5.3) within the prescribed period before the SV.
* Subject is currently a smoker or has used any tobacco products within 1 year or has a >10-pack/year smoking history (ie, the equivalent of smoking 1 pack per day per 10 years).
* Subject has any piercings of the tongue, lips, or mouth.
* Other criteria may apply, please contact the investigator for more information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time (AUC0-t) | Baseline, up to 24 hours
  At each treatment period
Maximum observed plasma drug concentration (Cmax) | Baseline, up to 24 hours
  At each treatment period

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time (AUC0-∞) | Baseline, up to 24 hours
  At each treatment period
Time to maximum observed plasma drug concentration (tmax) | Baseline, up to 24 hours
  At each treatment period
Terminal elimination half-life (t½) | Baseline, up to 24 hours
  At each treatment period
Summary of Participants with Adverse Events | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site, San Antonio, Texas, United States